CLINICAL TRIAL: NCT07280429
Title: A Study on Rehabilitation Study for Immune Checkpoint Inhibitors-Associated Myocarditis: A Randomized Controlled Trial
Brief Title: ICIAM Rehabilitation Program Study: A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Collaborators: Weifang Hospital of Traditional Chinese Medicine (Unknown); Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Jingyi Ren, Professor of medicine(Cardiology), Deputy Director of the Cardiology Department and Director of the Heart Failure Center, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023ZD0502805-02
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Immune Checkpoint Inhibitors Related Myocarditis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehab Arm (Experimental): The pharmacological rehabilitation protocol consists of oral administration of Shengxian Quyu Decoction. The traditional Chinese exercise rehabilitation protocol is designed following the FITT (Frequency, Intensity, Time, Type) principles of exercise therapy. Exercise modalities may include Baduanjin, with specific frequency, duration, and intensity tailored to each participant's actual condition. The total treatment period is 2 weeks.
  Interventions: Other: rehabilitation protocol
- Control Arm (No Intervention): The control arm received conventional treatment.

INTERVENTIONS:
Other: rehabilitation protocol — The intervention protocol comprised a pharmacological component (Shengxian Quyu therapy) and a traditional Chinese exercise rehabilitation component.The traditional Chinese exercise rehabilitation protocol is designed following the FITT (Frequency, Intensity, Time, Type) principles of exercise therapy. Exercise modalities may include Baduanjin, with specific frequency, duration, and intensity tailored to each participant's actual condition.
  Arms: Rehab Arm

SUMMARY:
Immunotherapy has become a cornerstone in oncology; however, managing its associated adverse events poses a significant clinical challenge. Cardiotoxicity represents a major concern, among which myocarditis accounts for a considerable proportion. This condition is characterized by poor prognosis, highly heterogeneous outcomes, and a high prevalence of persistent cardiac dysfunction after the acute phase. The dual impact of myocardial injury and underlying malignancy severely compromises patients' quality of life. Currently, it remains unclear whether implementing rehabilitation strategies for this patient population can mitigate the aforementioned challenges. Therefore, we designed a randomized controlled trial to evaluate the efficacy and safety of a structured rehabilitation program for convalescent patients with ICIAM.

DETAILED DESCRIPTION:
Eligible patients who are suitable for rehabilitation therapy and meet the TCM syndrome differentiation criteria of "Yangqi Deficiency with Internal Retention of Phlegm and Stasis" will be screened and undergo baseline assessments. Subsequently, they will be randomly assigned in a 1:1 ratio using block randomization to either the experimental group or the control group. The experimental group will receive a rehabilitation regimen consisting of Shengxian Quyu Decoction and specialized traditional Chinese exercise therapy, while the control group will receive conventional treatment only.The pharmacological rehabilitation intervention for the experimental group involves oral administration of Shengxian Quyu Decoction. The traditional exercise regimen is designed in accordance with the FITT principle (Frequency, Intensity, Time, Type) of exercise rehabilitation. Exercise modalities may include Baduanjin, with specific frequency, duration, and intensity tailored to individual patient conditions.The total rehabilitation period is 2 weeks. A follow-up assessment will be conducted at the end of the second week to document exercise adherence and evaluate physical examination findings, laboratory test results, TCM syndrome scores, quality of life, and Major Adverse Cardiovascular Events (MACE). Extended follow-up will continue through week 4 for MACE assessment.

ELIGIBILITY:
Inclusion Criteria:

* ①Aged 18 to 80 years, inclusive.②Malignancy confirmed by cytology or histopathology.③Diagnosis of ICIAM following ICI therapy.④Assessed by the Multidisciplinary Team for Immune-Related Adverse Events as clinically recovered and entering the rehabilitation.⑤Meet TCM syndrome differentiation criteria for "Yangqi Deficiency with Internal Retention of Phlegm and Stasis."⑥ KPS score > 60, with a life expectancy > 6 months.

Exclusion Criteria:

* ①Diagnosis of fulminant myocarditis or cardiac function of NYHA IV.②Clear evidence suggesting cardiac injury not attributable to ICIs.③Concurrent acute cardiovascular events or malignant arrhythmias.④Coexisting severe immune-related adverse events affecting other organ systems.⑤Associated severe systemic diseases, such as severe hepatic or renal insufficiency, or severe infection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
MACE | 2 weeks
  Cardiovascular Death, Cardiac Arrest, Cardiogenic Shock, High-Grade Atrioventricular Block
NT-proBNP/BNP levels | 2 weeks
  change in natriuretic peptide levels from baseline to Week 2
EQ-5D | 2 weeks
  Change in EQ-5D quality of life score

SECONDARY OUTCOMES:
MACE | 2 and 4 weeks
  Rates of individual MACE components

OTHER OUTCOMES:
Exercise adherence | 2 weeks
  Documenting patient exercise adherence

CONTACTS AND LOCATIONS:
Overall Officials: Jingyi Ren, Professor, Principal Investigator — China-Japan Friendship Hospital

IPD SHARING:
Plan to Share IPD: No